CLINICAL TRIAL: NCT04823104
Title: Optimizing Access to Care During Pregnancy in Rural Areas in a Perinatal Health
Brief Title: Optimizing Access to Care During Pregnancy in Rural Areas in a Perinatal Health Network
Acronym: OPTI'SOINS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to recruitment and implementation difficulties, the study was stopped prematurely
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREPS 2019 DEBOST-LEGRAND
Record Dates: First submitted 2021-03-23; First posted 2021-03-30 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy; Living in an Isolated Area
Keywords: Pregnancy; Home visitation; Isolated geographic area

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group with home visitation (Experimental): pregnant women who are included in this group will be assigned an intervention by home visitation for pregnancy follow-up
  Interventions: Other: Home visitation
- control group without home visitation (No Intervention): pregnant women will be free to choose their pregnancy follow-up without home visitation

INTERVENTIONS:
Other: Home visitation — Home visitation for pregnancy follow-up
  Arms: Intervention group with home visitation

SUMMARY:
Pregnant women who live in rural area have fewer prenatal consultations. It has been demonstrated that maternal and neonatal morbidity and mortality increase if time travel to a maternity ward is longer than 30 min.

Home visitation in isolated area may improve prenatal follow-up as it gives full access to women to health care professionals as well as biological and ultrasound exams without travelling.

Our aim is to assess the impact of home visitation on prenatal follow-up as compared to prenatal follow-up in maternity ward and in primary care.

Isolated areas will be randomized, for women living in areas included in the intervention group, home visitations will be planned for prenatal follow-up. Ultrasound screening as well as blood exams will be performed during home visitations. For women living in control areas, they will be free to choose prenatal follow-up modalities.

ELIGIBILITY:
Inclusion Criteria:

* At the first antenatal consultation, confirming the pregnancy.
* Pregnant women who live in an area of geographic vulnerability covered by a perinatal network
* The women must be informed about the study, understand, read, and speak French, and must be able to consent to participate in medical research

Exclusion Criteria:

* Pregnant women who live outside an area of geographic vulnerability covered by a perinatal network
* Women who give birth in a maternity ward outside Auvergne
* Women from another region giving birth in a maternity ward in Auvergne

Ages: 12 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
adequate pregnancy follow-up according to the French recommendations | 9 months
  number of consultations, In all, 8 consultations should take place in a pregnancy that goes to term
adequate pregnancy follow-up according to the French recommendations | 9 months
  number of ultrasound exams, Three systematic or screening ultrasound examinations, one per trimester, are recommended
adequate pregnancy follow-up according to the French recommendations | 9 months
  number of biological exams of recommended laboratory tests for antenatal care

SECONDARY OUTCOMES:
Adherence to antenatal care consultations of women | 9 months
  Adherence to the applicable French regulations concerning the term and number of consultations that must be performed until delivery
Adherence to antenatal care complementary exams of women by the mobile antenatal care clinic | 9 months
  The performance of all of the recommended ultrasounds at the recommended dates and all of the mandatory or recommended laboratory tests for antenatal care
adverse neonatal outcome | 9 months
  prematurity, in utero death, small or large for gestational age, transfer in intensive unit
adverse maternal outcome | 10 months
  gestational hypertension, preeclampsia, gestational diabetes, post-partum hemmorage, maternal death, transfer in intensive unit
economic analyse of the intervention | 24 months
  cost of equipment, human resources, balanced to income inherent to the project in accordance with the standards of cost budget accounting by insurance perspective.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, AURA, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Debost-Legrand A, Legrand G, Duclos-Medard J, Thomazet J, Pranal M, Langlois E, Mourgues C, Vendittelli F. Opti'care protocol: a randomised control trial to evaluate the impact of a mobile antenatal care clinic in isolated rural areas on prenatal follow-up. BMJ Open. 2023 Feb 16;13(2):e060337. doi: 10.1136/bmjopen-2021-060337. PMID 36797021